CLINICAL TRIAL: NCT04945993
Title: Assessment of Tooth Retention 10 Years After Root Canal Treatment With Endomethasone N: a Retro-prospective, National and Multicentre Clinical Study
Brief Title: Tooth Retention After Root Canal Treatment With Endomethasone N
Acronym: ENDO2021-02
Status: Active, not recruiting | Type: Observational
Sponsor: Septodont (Industry)
Responsible Party: Sponsor
Other Study IDs: ENDO-N
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Dental Root Canal Obturation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endomethasone N — Endomethasone N is a powder intended to be mixed extemporaneously with a eugenol-based liquid (i.e, Endomethasone Liquid) to obtain a permanent root canal sealer. After selection of dentists, they will screen consecutively and systematically eligible patients, will send them the Patient Information Letter and will enroll them in the clinical investigation if non opposition from the patient. Patient clinical data will be recorded in an electronic Case Report Form. Pseudonymized retro-alveolar radiographies at baseline consultation and at 5 and 10 years post-obturation consultations will be recorded in the e-CRF. These radiographies will be examined by 2 independent endodontists and the results of these examinations will be recorded in the e-CRF. Site data will be collected on a Site Questionnaire with Visual Analog Scales.

SUMMARY:
The aim of root canal treatment, or endodontic treatment, is to treat pulpal or periapical diseases and thus transform a pathological tooth into a healthy, asymptomatic and functional entity on the dental arch. The diagnosis of pulp pathology is based on the symptomatology described by the patient, on data from the clinical examination and tests performed as well as the radiographic examinations.

Different families of root canal sealers are used in endodontics: cements based on zinc oxide-eugenol (ZOE), resin-based materials, and calcium silicate-based cements. They provide a stable and hermetic sealing. The Septodont laboratory has developed and manufactured endomethasone N, a zinc oxide-eugenol root canal sealer.

The aim of this retro-prospective PMCF study is to collect long term clinical and safety data on root canal obturation after treatment or retreatment by Endomethasone N.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, > 18 years of age at the time of inclusion in the study
* Patient who had a non-surgical root canal treatment with Endomethasone N, in a context of an endodontic treatment, or retreatment, before 01-Mar-2016
* Having a documented patient follow-up visit (clinical examination and radiographic examination) at least 5 years after the endodontic treatment or retreatment with Endomethasone N
* Patient affiliated or beneficiary of a social security system
* Patient informed about the study and who confirm their non-opposition in participating in the study

Exclusion Criteria:

* History of malignant tumors in the 5 years prior to the root canal treatment
* Non-stabilized systemic disease during the month prior to the root canal treatment (diabetes, hypertension, thyroid disorders, etc.)
* Patient who developed a systemic pathology after the root canal treatment with Endomethasone N
* Patient who had endodontic treatment with Endomethasone N obturation on a wisdom tooth
* Patient whose tooth has suspected perforation during endodontic treatment
* Patient suffering from active non-stabilized periodontitis, untreated during endodontic treatment
* Patients participating in an interventional clinical trial at the time of root canal treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of root canal treatment.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Assessment of tooth functional retention | 10 years
  Rate of tooth functional retention after Root Canal Treatment with Endomethasone N

SECONDARY OUTCOMES:
Assessment of tooth functional retention | 5 years
  Rate of tooth functional retention after Root Canal Treatment with Endomethasone N.
Assessment of the tooth functional retention after Root Canal Treatment with Endomethasone N according to initial treatment or retreatment | 5 and 10 years
  Rate of tooth functional retention after Root Canal Treatment with Endomethasone N according to initial treatment or retreatment, on the basis of the same definition above
Assessment of the periapical healing | 5 and 10 years
  The periapical healing (success of obturation with Endomethasone N based on radiological criteria) at 5 and 10 years after Root Canal Treatment, will be evaluated in patients with retro-alveolar radiographs at the follow-up consultation (in parallel of the baseline consultation).
  The periapical healing is defined as follows:
  * a periapical status considered "normal" (PAI score <3) (See Appendix 2)
  * no resorption of the filling cement in the root, detectable on radiography
  * dense and homogeneous filling, limited to the canal,
  * a filling with the maintenance of the canal anatomy
The technical characteristics of the sealer Endomethasone N | 5 and 10 years
  The technical characteristics of the sealer Endomethasone N at 5 and 10 years after Root Canal Treatment "Not resorbable once hardened", "Not retractable over the years" and "Radiopaque" will be evaluated in patients with retro-alveolar radiographs at the follow-up consultation (in parallel of the baseline consultation). The technical characteristics are defined as follows:
  * no resorption of the filling cement in the root, detectable on radiography
  * dense and homogeneous filling, limited to the canal, with no apparent void along the root canal walls
  * a filling with the maintenance of the canal anatomy
The ease of use and insertion of Endomethasone N in the canal | 5 and 10 years
  The ease of use and insertion of Endomethasone N in the canal will be evaluated with the score obtained on the Visual Analog Scale: score from 0 (Not at all) to 10 (Certainly Yes).
The Investigator overall satisfaction of the experience with Endomethasone N | 5 and 10 years
  The Investigator overall satisfaction of the experience with Endomethasone N will be evaluated at 5 and 10 years after Root Canal Obturation with the score obtained on the Visual Analog Scale : score from 0 (Not at all) to 10 (Certainly Yes).
The immediate and long-term post-obturation adverse device effects | Immediately after root canal filling, and at long-term (i.e. 5 and 10 years)
  The immediate and long-term post-obturation adverse device effects will be evaluated with the list of adverse events immediately appearing after root canal filling and appearing at long-term (5 and 10 years) after root canal filling

CONTACTS AND LOCATIONS:
Overall Officials: Davy Aubeux, Dr, Study Director — Cabinet dentaire; Frank LEBRET, Dr, Principal Investigator — Cabinet dentaire; Vincent ROUBINET, Dr, Principal Investigator — Cabinet dentaire; Alain PHAM, Dr, Principal Investigator — Cabinet dentaire; Frederic JACOB, Principal Investigator — Cabinet dentaire
Locations (5):
- France (5):
  - Private dentist office - Dr PHAM, Athis-Mons
  - Private dentist office - Dr LEBRET, Dax
  - Private dentist office - Dr ROUBINET, Montélimar
  - Private dentist office - Dr AUBEUX, Saint-Herblain
  - Private dentist office - Dr JACOB, Valence

IPD SHARING:
Plan to Share IPD: Undecided